CLINICAL TRIAL: NCT03137407
Title: A Phase 2, Prospective, Randomized, Double-Blinded, Placebo-Controlled Trial of DaxibotulinumtoxinA for Injection for the Management of Plantar Fasciitis
Brief Title: Phase 2 DaxibotulinumtoxinA for Injection for the Management of Plantar Fasciitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Revance Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1720201
Record Dates: First submitted 2017-04-27; First posted 2017-05-02 (Actual); Results first posted 2023-08-28 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-08

CONDITIONS: Plantar Fasciitis
Keywords: heel pain
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DAXI 240 U (Experimental): DaxibotulinumtoxinA for injection for the treatment of plantar fasciitis (PF) with 240 U
  Interventions: Biological: Botulinum Toxins, Type A
- Placebo (Placebo Comparator): Placebo Intramuscular Injection
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Botulinum Toxins, Type A — Intramuscular injection
  Other Names: DaxibotulinumtoxinA
  Arms: DAXI 240 U
Biological: Placebo — Intramuscular injection
  Arms: Placebo

SUMMARY:
The specific aim of the study is to compare the safety and efficacy of a single administration of DaxibotulinumtoxinA for Injection versus placebo for managing plantar fasciitis.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent, including authorization to release health information
* Male or female subjects 18 to 65 years of age with diagnosis of plantar fasciitis
* Persistent heel pain for more than three months
* Women of child bearing potential must have negative pregnancy test at Screening and Injection Visits and must use an effective method of birth control during the course of the study

Exclusion Criteria:

* Previous surgery on the midfoot or hindfoot
* Neuromuscular disease
* Systemic muscle weakness
* Planning a pregnancy during the study
* Current enrollment in an investigational drug or device study or participation in such a study within the last 30 days prior to first visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-02-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Village Podiatry Centers, Duluth, Georgia
  - Weil Foot and Ankle Institute, Des Plaines, Illinois
  - Kansas City Bone & Joint Clinic, Overland Park, Kansas
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Element Research Group, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo group
Period: Overall Study
Arm/Group | DAXI 240 U | Placebo
Started | 30 | 29
Completed | 26 | 23
Not Completed | 4 | 6

BASELINE CHARACTERISTICS:
Population: 59 subjects were enrolled. Subjects were assigned to study if they met all inclusion and none of the exclusion criteria. All subjects enrolled were randomized and received study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | DAXI 240 U | Placebo | Total
Number analyzed (Participants) | 30 | 29 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (9.17) | 46.9 (9.61) | 46.9 (9.31)
Age, Customized [Count of Participants; unit: Participants]
  <30 | 1 | 1 | 2
  30 - <40 | 7 | 6 | 13
  40 - <50 | 8 | 11 | 19
  50 - <60 | 11 | 7 | 18
  >=60 | 3 | 4 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 22 | 42
  Male | 10 | 7 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 25 | 20 | 45
  Black/African American | 5 | 8 | 13
  Mixed Race/Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Week 8 in the Visual Analog Scale (VAS) for Pain for the Foot
Description: The primary efficacy endpoint, as identified in the Statistical Analysis Plan (SAP) was the change from baseline in the visual analog scale (VAS) for pain for the affected foot at Week 8.
  The outcome was measured by means of a 100 mm VAS (0= no pain, 100= maximum pain) and higher reduction from baseline VAS pain scores means a better outcome.
Time Frame: Week 8
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- DaxibotulinumtoxinA 240 Units: Botulinum Toxins, Type A Intramuscular Injection
  Botulinum Toxins, Type A: Intramuscular injection
Arm/Group | DaxibotulinumtoxinA 240 Units | Placebo
Number analyzed (Participants) | 30 | 29
score on a scale | -41.6 (30.04) | -39.3 (32.54)

2. Secondary Outcome: Change From Baseline in Foot Pain as Measured by the Visual Analog Scale (VAS) Through Week 16
Description: Reduction in foot pain was assessed as the change from baseline in the Visual Analog Scale (VAS) at weeks 1, 2, 4, 8, and 16. The outcome was measured by means of a 100 mm VAS (0= no pain, 100= maximum pain) and higher reduction from baseline VAS pain scores means a better outcome.
Time Frame: Weeks 1, 2, 4, 8, and 16
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DAXI 240 U | Placebo
Number analyzed (Participants) | 30 | 29
score on a scale
  Week 1 | -27.4 (28.92) | -21.6 (26.79)
  Week 2 | -31.6 (29.97) | -29.6 (27.33)
  Week 4 | -37.9 (27.15) | -31.4 (28.96)
  Week 8 | -41.6 (30.04) | -39.3 (32.54)
  Week 16 | -44.7 (32.82) | -46.3 (30.40)

3. Secondary Outcome: Change From Baseline Through Week 16 for the American Orthopaedic Foot and Ankle Score (AOFAS)
Description: The American Orthopaedic Foot and Ankle Score (AOFAS) measures foot and ankle conditions in 3 categories, pain, function, and alignment. The scale includes 9 items and the total score ranges from a minimum of 0 to a maximum of 100, with higher scores indicating a better outcome.
Time Frame: Weeks 1, 2, 4, 8, and 16
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DAXI 240 U | Placebo
Number analyzed (Participants) | 30 | 29
score on a scale
  Week 1 | 12.4 (17.56) | 15.5 (16.85)
  Week 2 | 14.3 (20.32) | 18.5 (16.85)
  Week 4 | 19.4 (22.76) | 21.2 (20.06)
  Week 8 | 20.4 (23.64) | 23.6 (24.88)
  Week 16 | 25.7 (23.41) | 23.1 (24.05)

4. Secondary Outcome: Change From Baseline Through Week 16 for the Foot and Ankle Disability Index
Description: The Foot and Ankle Disability Index is a 26 item questionnaire that measures disability and measures a total value minimum of 0 to a maximum of 104, with higher scores indicating greater disability.
Time Frame: Weeks 1, 2, 4, 8, and 16
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DAXI 240 U | Placebo
Number analyzed (Participants) | 30 | 29
score on a scale
  Week 1 | 9.1 (16.63) | 14.5 (14.87)
  Week 2 | 10.4 (16.93) | 16.5 (14.12)
  Week 4 | 16.4 (20.66) | 19.3 (14.21)
  Week 8 | 19.1 (20.98) | 19.7 (15.71)
  Week 16 | 21.7 (22.60) | 23.2 (17.86)

ADVERSE EVENTS:
Time Frame: Up to week 16
Description: Adverse events are summarized in terms of incidence of Treatment Emergent Adverse Events. Safety was assessed on all randomized (59) patients who received study treatment and were assessed for safety at least once after baseline
Arm/Group | DAXI 240 U | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/29
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/29
Other Adverse Events (participants affected / at risk) | 20/30 | 16/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DAXI 240 U (N=30) | Placebo (N=29)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DAXI 240 U (N=30) | Placebo (N=29)
Atrioventricular block first degree (Cardiac disorders) | 0 | 2
Injection Site Hemorrhage (General disorders) | 3 | 2
Injection Site Pain (General disorders) | 6 | 6
Injection site bruising (General disorders) | 2 | 1
Injection site edema (General disorders) | 0 | 2
Injection site erythema (General disorders) | 0 | 2
Paronychia (Infections and infestations) | 2 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 3
Headache (Nervous system disorders) | 0 | 2
Hypoaesthesia (Nervous system disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study Center and/or Investigator shall submit to Revance a copy of the proposed publication at least sixty (60) days prior to the submission thereof for publication or disclosure to a third party: (i)to provide Revance with the opportunity to review and comment on the contents thereof, (ii)to identify any Confidential Information to be deleted from the proposed publication or disclosure, and (iii)or delay the publication or disclosure 90 days to allow Revance to pursue patent protections.

DOCUMENTS (2):
  • Study Protocol (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/07/NCT03137407/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/07/NCT03137407/SAP_001.pdf